CLINICAL TRIAL: NCT03440346
Title: Biomarker Research in ADHD: the Impact of Nutrition (BRAIN). An Open-label Trial to Investigate the Mechanisms Underlying the Effects of a Few-foods Diet on ADHD Symptoms in Children
Brief Title: Biomarker Research in ADHD: the Impact of Nutrition
Acronym: BRAIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Collaborators: ADHD Research Centre (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NL63851.081.17
Record Dates: First submitted 2018-01-19; First posted 2018-02-22 (Actual); Last update posted 2019-07-01 (Actual); Status verified 2019-06

CONDITIONS: Attention Deficit-Hyperactivity Disorder
Keywords: Attention Deficit Hyperactivity Disorder; ADHD; child; human; diet; few-foods diet; brain; gut; microbiota
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Few-foods diet intervention (Experimental)
  Interventions: Other: Few-foods diet

INTERVENTIONS:
Other: Few-foods diet — The few-foods diet (FFD) is followed for 5-weeks preceded by a 1-week transition period during which the child's eating pattern will be gradually adjusted. The diet consists of rice, meat (turkey and lamb), a range of vegetables, pear, rice milk with added calcium and water, and is complemented with foods such as potatoes, fruits, corn, some sweets and wheat, which are allowed in small quantities only. Normal quantities of vegetables, rice and meat are allowed every day. If necessary the diet will be adjusted to avoid foods that the child dislikes or has cravings for. If the child does not respond to the initial FFD, i.e. no change in behaviour after the first two weeks, interim adjustments to the FFD will be made in consultation with the parents.
  Other Names: Restricted Elimination Diet

SUMMARY:
Attention deficit hyperactivity disorder (ADHD) is the most common childhood behavioural disorder, causing significant impediment to a child's development. The exact aetiology of ADHD is still unknown. It is a complex disorder with numerous contributing (epi)genetic and environmental factors. Currently, treatment predominantly consists of behavioural and pharmacological therapy. However, medication use is associated with several side effects and concerns about long-term effects and efficacy exist. Therefore, there is considerable interest in the development of alternative treatment options.

Double-blind research investigating the effect of a few-foods diet (FFD) has demonstrated large improvements in ADHD symptoms. However, following an FFD requires great effort of both the child and parents. To make this treatment easier or potentially obsolete, it is important to understand how and in which children an FFD affects ADHD symptoms.

The investigators hypothesise that an FFD affects brain function and behaviour, including ADHD symptoms, via the complex network of communication between the microbiota, gut and brain, i.e. the MGB axis. The aim of this study is to identify potential mechanism(s) underlying the impact of an FFD on ADHD symptoms and to identify biomarkers that predict the response to the FFD.

100 boys with ADHD will follow the FFD for 5 weeks. After inclusion, all participants will start with a baseline period, during which they will maintain their regular diet. The baseline period ends at the end of week 2. Thereafter, participants will follow a 5-week FFD, preceded by a 1-week transition period. The FFD period ends at the end of week 8.

At the end of the baseline period (i.e. at the end of week 2) and at the end of the FFD (i.e. at the end of week 8), fMRI scans will be made, blood and buccal saliva will be collected, and stool and urine will be handed in. Children will do computer tasks and parents will complete questionnaires to monitor ADHD and physical complaints. All samples will be analysed by researchers blinded to behavioural responses to the FFD. To assess the impact of the FFD on brain function and the MGB axis, associations between ADHD behavioural changes and changes in other primary and secondary study outcomes will be analysed.

This study may lead to the identification of biomarkers that can predict the response to an FFD. Understanding which changes - induced by an FFD - lead to improvements in ADHD symptoms may provide new avenues for developing treatments. Ultimately, the findings may enable personalised intervention strategies based on an individuals' configuration of the MGB axis.

ELIGIBILITY:
Inclusion Criteria:

* Meeting DSM-IV ADHD criteria
* Male
* Aged 8 up to and including 10 years
* Right-handed
* Available to visit Wageningen University for 4 sessions (i.e. intake, screening, T1 and T2), of which 3 sessions including the child (screening, T1, T2)
* Upon study start, fully understanding and agreeing to the study objectives and having dated and signed an informed consent to participate in the study, including permission that material will be used or archived for (epi)genetic testing
* Willing to be informed about chance-findings that may have implications for the health of the child or his family, and approving of reporting this to the child's medical specialist or family's general physician.
* If the child uses "over the counter" medication, e.g. laxatives, melatonin for sleeping problems or hay fever medication, parents are asked to share the information leaflet, and if necessary participants are asked to change to alternatives that are free of additives that may affect ADHD, e.g. laxatives free of artificial sweeteners, sugar and cacao.

Exclusion Criteria:

* Diagnosis Autism Spectrum Disorder
* Diagnosis Developmental Coordination Disorder
* Premature birth (< 36 weeks) and/or oxygen deprivation during birth
* Diagnosed chronic gastrointestinal disorder, i.e. inflammatory bowel disease, irritable bowel syndrome, celiac disease, non-celiac gluten-intolerance (gluten-sensitivity) or lactose-intolerance
* Auto-immune disorder (e.g. diabetes mellitus type 1)
* Vegetarian/vegan
* Diagnosis dyslexia and/or dyscalculia
* IQ < 85
* Following behavioural therapy
* Use of ADHD medication
* Use of systemic antibiotics, antifungals, antivirals or antiparasitics in the past six months
* Insufficient command of the Dutch language by either parents or child that may affect understanding and execution of study and dietary instructions
* Family circumstances that may compromise following or completion of the diet, including but not limited to family relational problems
* Having a contra-indication to MRI scanning (including, but not limited to): pacemakers and defibrillators, intraorbital or intraocular metallic fragments, ferromagnetic implants, claustrophobia.
* Two weeks prior to the start of the study, dietary supplements (e.g. antioxidants, minerals, vitamins) or pro- or prebiotics use has to be stopped.

Ages: 8 Years to 10 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2018-02-19 (Actual); Primary Completion 2019-06-21 (Actual); Study Completion 2019-06-21 (Actual)

PRIMARY OUTCOMES:
Change in neural activation patterns during execution of tasks | Before and at the end of the FFD intervention (i.e. at the end of week 2 and at the end of week 8)
  Using fMRI, blood oxygen-level-dependent (BOLD) signal changes will be measured whilst performing cognitive tasks that assess inhibitory control and selective attention, i.e. a stop-signal task (response inhibition) and a Flanker task (response conflict and associated error monitoring). fMRI BOLD responses will be assessed between variable task-elements and performance. Region of interest (ROI; anatomically defined regions in the brain) analyses of the BOLD responses will be performed.
Change in peripheral blood metabolite concentrations | Before and at the end of the FFD intervention (i.e. at the end of week 2 and at the end of week 8)
  Global metabolite profiles will be examined in plasma (or alternatively serum) obtained from whole blood using mass-spectrometry profiling. Phenylalanine and tyrosine plasma levels represent primary outcomes.
Change in functional composition of the gut microbiota | Before and at the end of the FFD intervention (i.e. at the end of week 2 and at the end of week 8)
  Metagenome profiling will be performed on stool samples, leveraging Illumina next-generation sequencing technology. Sequence read data will be used for abundance profiling of microbiota genes that encode enzymes directly involved in the production or degradation of the dopamine and noradrenaline precursors phenylalanine and tyrosine.
Change in ADHD symptom scores | Before and at the end of the FFD intervention (i.e. at the end of week 2 and at the end of week 8)
  ADHD symptoms will be scored using the 18-item ADHD rating scale, which is based on the Diagnostic and Statistical Manual of Mental Disorders (DSM)-IV and consists of 9 items that assess inattention and 9 items that focus on hyperactivity and impulsivity.

SECONDARY OUTCOMES:
Change in whole brain neural activation patterns during the execution of tasks | Before and at the end of the FFD intervention (i.e. at the end of week 2 and at the end of week 8)
  fMRI BOLD responses, assessed between variable task-elements, will be explored using whole brain imaging analyses.
Change in whole brain functional connectivity at rest | Before and at the end of the FFD intervention (i.e. at the end of week 2 and at the end of week 8)
  A resting-state fMRI scan will be performed to analyse the networks of brain structures that are active during the resting-state.
Change in taxonomic and functional composition of the gut microbiota | Before and at the end of the FFD intervention (i.e. at the end of week 2 and at the end of week 8)
  Stool metagenome and/or 16S ribosomal ribonucleic acid (rRNA) gene profiling will be performed using Illumina sequencing. Metagenome data will be used to determine the taxonomic and functional composition of the gut microbiota.
Change in metabolite profiles | Before and at the end of the FFD intervention (i.e. at the end of week 2 and at the end of week 8)
  Global metabolite profiles will be examined in plasma (or alternatively serum) obtained from whole blood, urine and optionally in stool using mass-spectrometry profiling.
Change in peripheral blood cell gene expression profiles | Before and at the end of the FFD intervention (i.e. at the end of week 2 and at the end of week 8)
  Peripheral blood mononuclear cells will be isolated from fasting blood samples and gene expression profiles will either be determined using Affymetrix gene expression arrays or by RNA-sequencing.
Change in a panel of peripheral blood protein biomarkers related to immune, metabolic and neurological status | Before and at the end of the FFD intervention (i.e. at the end of week 2 and at the end of week 8)
  A large panel of proteins will be profiled using quantitative immunoassays or proteomics on blood plasma or serum.
DNA genotype | Before the FFD diet intervention (i.e. at the end of week 2)
  Genotyping will be conducted using a microarray platform on DNA isolated from buccal cells or on DNA isolated from whole blood.
Change in DNA methylation profiles | Before and at the end of the FFD intervention (i.e. at the end of week 2 and at the end of week 8)
  Genome-wide profiling of DNA methylation status will be conducted using the Illumina Infinium MethylationEPIC beadchip microarray platform in DNA isolated from buccal cells or alternatively on DNA isolated from whole blood.
Change in executive function | Before and at the end of the FFD intervention (i.e. at the end of week 2 and at the end of week 8)
  Executive functioning will be measured using a continuous performance test that assesses executive functions such as sustained attention and behavioural inhibition.
Change in ADHD symptoms | Before and at the end of the FFD intervention (i.e. at the end of week 2 and at the end of week 8)
  Change will be scored using the Abbreviated Conners' scale
Change in oppositional defiant disorder symptoms | Before and at the end of the FFD intervention (i.e. at the end of week 2 and at the end of week 8)
  Change will be scored using a validated questionnaire.
Change in social behavioural problems | Before and at the end of the FFD intervention (i.e. at the end of week 2 and at the end of week 8)
  Change will be scored using the children's social and behavioural questionnaire.
Change in physical complaints | Before and at the end of the FFD intervention (i.e. at the end of week 2 and at the end of week 8)
  Change will be scored using a validated questionnaire.
Change in stool frequency | Before and at the end of the FFD intervention (i.e. at the end of week 2 and at the end of week 8)
  The child will record the frequency of defaecations for one week.
Change in stool type | Before and at the end of the FFD intervention (i.e. at the end of week 2 and at the end of week 8)
  The child will type each stool using the modified Bristol stool scale form for children, which comprises 5 stool form types described and depicted in drawings.

OTHER OUTCOMES:
IQ-score | At the screening session, prior to inclusion of participant in the study
  If no intelligence quotient (IQ) test has been conducted in the past year, an abbreviated form of the Wechsler Intelligence Scale III IQ test will be conducted.
Change in taxonomic and functional composition of the gut microbiota | Prior to the screening (i.e. week 0) and after the baseline period (i.e. at the end of week 2)
  Stool metagenome and/or 16S rRNA gene profiling will be performed using Illumina sequencing. Metagenome data will be used to determine the taxonomic and functional composition of the gut microbiota. The change in gut microbiota composition will be assessed between stools sampled prior to the screening and after the baseline period (i.e. before the start of the FFD intervention).

CONTACTS AND LOCATIONS:
Overall Officials: Michiel Kleerebezem, Prof. dr., Principal Investigator — Wageningen University
Locations (1):
- Wageningen University, Wageningen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pelsser LM, Frankena K, Toorman J, Savelkoul HF, Dubois AE, Pereira RR, Haagen TA, Rommelse NN, Buitelaar JK. Effects of a restricted elimination diet on the behaviour of children with attention-deficit hyperactivity disorder (INCA study): a randomised controlled trial. Lancet. 2011 Feb 5;377(9764):494-503. doi: 10.1016/S0140-6736(10)62227-1. PMID 21296237
- [Background] Pelsser LM, Frankena K, Toorman J, Rodrigues Pereira R. Diet and ADHD, Reviewing the Evidence: A Systematic Review of Meta-Analyses of Double-Blind Placebo-Controlled Trials Evaluating the Efficacy of Diet Interventions on the Behavior of Children with ADHD. PLoS One. 2017 Jan 25;12(1):e0169277. doi: 10.1371/journal.pone.0169277. eCollection 2017. PMID 28121994
- [Derived] Stobernack T, de Vries SPW, Rodrigues Pereira R, Pelsser LM, Ter Braak CJF, Aarts E, van Baarlen P, Kleerebezem M, Frankena K, Hontelez S. Biomarker Research in ADHD: the Impact of Nutrition (BRAIN) - study protocol of an open-label trial to investigate the mechanisms underlying the effects of a few-foods diet on ADHD symptoms in children. BMJ Open. 2019 Nov 5;9(11):e029422. doi: 10.1136/bmjopen-2019-029422. PMID 31694844
- See also: BRAIN-study website — http://www.brain-studie.nl